CLINICAL TRIAL: NCT03579017
Title: Cognitive Impairment in ALS: Screening Tools, Experiences and Prognosis
Brief Title: Edinburgh Cognitive and Behavioural Amyotrophic Lateral Sclerosis Screen in Norway: A Validation Study
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Western Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/3166
Record Dates: First submitted 2018-06-01; First posted 2018-07-06 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Amyotrophic Lateral Sclerosis; Cognitive Impairment
Keywords: Amyotrophic lateral sclerosis; Cognitive; Screening; Validation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with ALS: Patients with ALS will be tested by two independent testers with the ECAS-N at 4 months (baseline) and 8 months (follow-up), and the MoCA at 4 months (baseline) by one tester
  Interventions: Diagnostic Test: ECAS-N; Diagnostic Test: MoCA
- Healthy controls: Persons with no cognitive impairment will be tested with the ECAS-N once, by one tester
  Interventions: Diagnostic Test: ECAS-N
- Controls with dementia: Persons with cognitive impairment due to other disorders will be tested with the ECAS-N once, by one tester
  Interventions: Diagnostic Test: ECAS-N

INTERVENTIONS:
Diagnostic Test: ECAS-N — All participants included will be tested with the ECAS-N
  Other Names: Edinburgh cognitive and behavioral ALS screen (Norwegian)
Diagnostic Test: MoCA — All included patients With ALS will be tested With the MoCA
  Other Names: Montreal cognitive assessment (MoCA)
  Groups: Patients with ALS

SUMMARY:
Cognitive impairment is present in about 30-50% of the patients with amyotrophic lateral sclerosis (ALS). Suitable screening tools are available, but none of these are evaluated in a Norwegian population.

DETAILED DESCRIPTION:
Screening of cognitive and behavioral impairment is a distinct recommendation in ALS-specific health-care. Thus, a rapid screening tool valid for use in Norway is urgent. However, cognitive assessment for patients with ALS can be difficult due to the complexity of cognitive impairment, as well as motor challenges with writing, drawing and speaking. Therefore, only ALS-specific, multi domain screening instruments with integrated behavioral sections should be used. Internationally, the Edinburgh cognitive and behavioral amyotrophic lateral sclerosis screen (ECAS), is recommended for the purpose. Besides being quick and easy to administer, the ECAS is shown to be sensitive and have high specificity to ALS-specific dysfunction and behavioral changes. The introduction of ECAS has probably contributed to a more nuanced picture of cognitive impairment in ALS than previously assumed. Therefore the ECAS has been translated and culturally adapted into Norwegian (ECAS-N). Based on scores from healthy people, Norwegian age- and educational-adjusted norms for verbal fluency (n=277) and cut-off-scores (n=85) for abnormal findings are established. However, further investigation of psychometric properties of the ECAS-N is needed. The objectives of the study are: 1. To investigate if the ECAS-N reflect cognitive impairment (internal consistency), and is robust to measurement errors due to different times of testing (test-retest reliability) and different raters (interrater reliability) 2. To investigate if the ECAS-N can be used to distinguish between people with ALS-specific cognitive impairment, and those who do not have cognitive impairment, and those who have cognitive impairment due to other disorders (construct validity).

ELIGIBILITY:
Inclusion Criteria:

* voluntary informed consent
* native Norwegian speaker
* aged between 35 and 85 years old (only for Controls)

Exclusion Criteria:

* great difficulties in writing og Reading
* comorbid Medical history
* neurological disorders others than ALS
* psychiatric history of importance to cognitive function

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who fulfill the inclution criteria and attending to the ALS-unit at HUH, St.Olavs Hospital, Hospital of Southern Norway or Namsos Hospital, within 4 months after being diagnosed With ALS.
  Healthy People and patients with dementia will constitute Control groups
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Edinburgh cognitive and behavioural amyotrophic lateral sclerosis screen - Norwegian Version (ECAS-N) | 4 months
  We will use the ALS-specific sub-score (minimum score = 0, maximum score = 100), the ALS non-specific sub-score (minimum score = 0, maximum score = 36), a summed total ECAS-N score (minimum score =0, maximum score =136), the sub score of behavioural changes (minimum score = 0, maximum score = 10) and the sub score of psychotic change (minimum score = 0, maximum score = 3). A dichotomized cut-off scores for normality will also be used for the ALS-specific cut-off score of 65 or over, the non ALS-specific cut-off score of 24 or over and the total ECAS-N cut-off score of 92 or over. For the ALS-specific scores, non ALS-specific scores and total ECAS-N scores, high scores indicate less problems than low scores. For the sub score of behavioural change and the sub score of psychotic change, high scores indicate more problems than low scores.

SECONDARY OUTCOMES:
Montreal cognitive assessment (MoCA) - Norwegian version | 4 months
  We will use the total MoCA score (minimum score = 0, maximum score = 30) and a dichotomized cut-off score for normality of 26 or over. High scores indicate less problems than low scores
Change from 4 months Edinburgh cognitive and behavioural amyotrophic lateral sclerosis screen - Norwegian Version (ECAS-N) at 8 months | 8 months
  We will use the changed ALS-specific sub-score (minimum score = 0, maximum score = 100), the changed ALS non-specific sub-score (minimum score = 0, maximum score = 36), a changed summed total ECAS-N score (minimum score =0, maximum score =136), the changed sub score of behavioural changes (minimum score = 0, maximum score = 10) and the changed sub score of psychotic change (minimum score = 0, maximum score = 3). A changed dichotomized cut-off scores for normality will also be used for the ALS-specific cut-off score of 65 or over, the non ALS-specific cut-off score of 24 or over and the total ECAS-N cut-off score of 92 or over. For the ALS-specific scores, non ALS-specific scores and total ECAS-N scores, high scores indicate less problems than low scores. For the sub score of behavioural change and the sub score of psychotic change, high scores indicate more problems than low scores.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Taule, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway